CLINICAL TRIAL: NCT02598869
Title: Posterior Subtenon Versus Intravitreal Injection of Triamcinolone Acetonide for Treatment of Uveitic Cystoid Macular Edema (CME)
Brief Title: Posterior Subtenon Versus Intravitreal Injection of Triamcinolone Acetonide for Treatment of Uveitic Cystoid Macular Edema
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Phoebe Lin, MD,PhD, Assistant professor of Ophthalmology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00011584
Record Dates: First submitted 2015-08-31; First posted 2015-11-06 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Uveitis; Cystoid Macular Edema
Keywords: Triamcinolone acetonide
MeSH Terms: conditions — Uveitis; Macular Edema | interventions — Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravitreal triamcinolone (Active Comparator): subjects will receive intravitreal injection of 2mg /0.05 ml of preservative free triamcinolone acetonide ( otherwise known as triesence)
  Interventions: Drug: Triamcinolone Acetonide
- posterior subtenon triamcinolone (Active Comparator): subjects will receive posterior subtenon injection of 40mg /1 ml of preserved triamcinolone acetonide ( otherwise known as kenalog)
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — injection of triamcinolone acetonide
  Other Names: triesence; kenalog

SUMMARY:
Macular edema is the most common sight threatening complication of uveitis which can lead to permanent loss of central vision. Triamcinolone acetonide ( the study drug)injection for treatment of cystoid macular edema(CME) is well established. The purpose of this study is to compare the safety and efficacy of injecting the study drug inside the eye(intravitreal injection) and behind the eye(subtenon injection)

DETAILED DESCRIPTION:
The study is randomized interventional non inferiority study that will enroll 30 adults aged 18 or older with the diagnosis of cystoid macular edema secondary to non-infectious uveitis. Potential subjects will be recruited from the retina and uveitis clinics at the Casey Eye Institute, Oregon health and science University(OHSU). Potential recruits will be asked to sign and date the informed consent and a copy will be given to subject prior to any study procedure. Subjects will have a screening visit before the injection procedure so that the study doctor can decide if they meet the criteria to be in the study. This study requires 6 visits to the clinic and will take 6 months to complete. During the screening visit, medical/ surgical/ ocular history and will be collected from the subject and medical records. Laboratory tests will be performed to rule out infectious uveitis if the subject has not already had infectious types of uveitis ruled out since the time of diagnosis of uveitis. Urine collection for pregnancy test for females of childbearing potential will be done. Examination of subjects will include measurement of visual acuity, examination of the front and back part of the eye, measurement of the eye pressure . A scan of the retina will be obtained by spectral domain optical coherence tomography (SD-OCT). During the injection visit, history, examination, and pregnancy tests will be repeated in addition to receiving the injection. Subjects will be randomized to either injecting the study drug by intravitreal or subtenon routes. Examination after injection will be performed to rule out immediate complications. Then subjects will have 4 follow-up visits (2 weeks, 1 month, 3 months and 6 months). During each visit, subjects will be asked about adverse events, concomitant medications, how their eyes feel in addition to obtaining a clinical examination and OCT.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female at least 18 years of age at the time of consent
* One or both eyes having CME associated with non-infectious uveitis
* Subject has the ability to understand and sign the Informed Consent Form
* Subject is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Allergy to triamcinolone acetonide
* History of any type of non-infectious uveitis without macular edema
* Vitreous hemorrhage
* Uveitis with infectious etiology
* CME due to non-uveitis causes
* Previous viral retinitis or uveitis
* Toxoplasmosis scar in study eye or scar related to viral retinitis
* Media opacity interfering with optical coherence tomography (OCT) or evaluation of the retina and vitreous
* Patient may not have had prior treatment for CME within the past 3 months including anti-VEGF (vascular endothelial growth factor), periocular or intravitreal steroid
* Pregnant or nursing women; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception
* Subjects unwilling to comply with the study protocol or who are likely to be lost to follow-up within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2016-05-15 (Actual); Study Completion 2016-05-15 (Actual)

PRIMARY OUTCOMES:
Mean change in best corrected visual acuity( BCVA) | at 1,3 and 6 months after intervention
  Best corrected visual acuity will be assessed using the Snellen chart

SECONDARY OUTCOMES:
Change in central macular thickness in micrometers | at 1,3 and 6 months after intervention
  A spectral domain optical coherence tomography device will be used to capture central macular thickness
Percentage of eyes that develop side effects | at 1,3 and 6 months after intervention

REFERENCES:
- [Background] Guex-Crosier Y. The pathogenesis and clinical presentation of macular edema in inflammatory diseases. Doc Ophthalmol. 1999;97(3-4):297-309. doi: 10.1023/a:1002130005227. PMID 10896343
- [Background] Sivaprasad S, McCluskey P, Lightman S. Intravitreal steroids in the management of macular oedema. Acta Ophthalmol Scand. 2006 Dec;84(6):722-33. doi: 10.1111/j.1600-0420.2006.00698.x. PMID 17083528
- [Background] Leder HA, Jabs DA, Galor A, Dunn JP, Thorne JE. Periocular triamcinolone acetonide injections for cystoid macular edema complicating noninfectious uveitis. Am J Ophthalmol. 2011 Sep;152(3):441-448.e2. doi: 10.1016/j.ajo.2011.02.009. Epub 2011 Jun 8. PMID 21652023